CLINICAL TRIAL: NCT00465335
Title: Multi-Detector Computer Tomography(MDCT)in Patients With Equivocal/Intermediate Post Test Probability of Coronary Artery Disease
Brief Title: Usefulness of Coronary CT Angiography in Patients With Inconclusive Stress Test Results
Acronym: IMPACCT
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Other Study IDs: 2005-135 IMPACCT
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Angiography; Coronary Disease
Keywords: computed tomography; stress test; equivocal; catheterization
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the usefulness of performing a "cat scan" of the heart arteries in patients (without a known history of heart disease) seen by their physician for chest pain. We plan to evaluate this test in patients who have already undergone stress testing. On occasion, stress test results are equivocal or suspected to be inaccurate. In these cases, depending on the overall clinical suspicion of coronary artery disease, physicians may recommend cardiac catheterization to determine whether or not patients have blockages in their heart's arteries. We plan to evaluate whether a Cat Scan of the heart arteries will provide your physician with important information to assist in this decision. If the results of this test are normal, the patient may not require a heart catheterization; alternatively, if the test is abnormal, a physician may proceed with catheterization after review of the data. There will 200 patients enrolled into the study. All patients will be followed by their usual cardiologist, and all decisions will be made by their cardiologist.

Computed tomography (CT; "cat scan") is an x-ray test routinely used for diagnostic purposes. Cardiac computed tomography using the newer generation multislice CT (MSCT) scanners is an improved way of using CT scanning techniques to look at the heart and blood vessels of the body. The images of the coronary arteries obtained by MSCT scanners (during a 5-10 minute procedure) are highly accurate, when compared to the conventional invasive cardiac catheterization procedure. This procedure will provide a calculation of a coronary artery calcium score as well as an accurate depiction of the coronary anatomy. The accuracy of this test is similar to that achieved with traditional stress test imaging, but has some inherent advantages over this traditional stress testing. Therefore, we believe that in patients with intermediate, inconclusive, or suspected inaccurate stress tests, MSCT of the coronary arteries may provide helpful information to your physician to help guide their decision regarding the need (or lack of) for possible invasive cardiac catheterization. This procedure is considered an ideal "screening test" to exclude the presence of coronary artery disease in patients with suspected coronary artery disease.

On the day of your procedure, the patient will be given intravenous ("IV dye") contrast during their Cat Scan. We will also draw a blood sample to assess your kidney function and/or pregnancy status (if necessary). The contrast is what creates the pictures of one's arteries. The intravenous contrast used is the same dye as that used for routine cat scans of other parts of the body, as well as for cardiac catheterization. Prior to the Scan patients may be prescribed a medicine called a beta blocker The beta blocker typically used is called Atenolol. This medication slows your heart rate and is one that is commonly used to treat high blood pressure. Dosing will be based upon your current medications and vital signs. If a patient's heart rate is greater than 60 beats per minute an intravenous beta-blocker may be given to optimize their heart images. Patient's will have to hold your breath twice, for up to 30 seconds each time. The imaging part of the test takes about 10 minutes. Patient's will be observed after the test for about 20 minutes, followed by discharge home. Physicians will called with the patient's results of the study, and they will contact their patient's regarding the results, as well as the "next step." If a patient is a diabetic (taking metformin/glucophage), we will request a follow up (the next day) kidney test. Patient's will also will be called at 3 months to asked a few brief questions regarding your health (any recent hospitalizations, any new medical illnesses, any follow up heart testing, etc.)

DETAILED DESCRIPTION:
The purpose of this observational study is to prospectively evaluate the impact of multi detector CT angiography (MDCT) in patients with equivocal/intermediate post exercise stress test probability of coronary artery disease.

The primary objective are to:

1. Evaluate the diagnostic and prognostic performance of MDCT in patients with equivocal/ intermediate post test probability of CAD and
2. Evaluate the accuracy of MDCT in prediction of 30 day major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Patient with Chest Pain or other symptoms suggestive of Coronary Artery Diseae
* Stress ECG, Stress Echo, or Stress Nuclear in past 6 months.
* Equivocal test results or discordant clinical/stress information
* Able to provide consent

Exclusion Criteria:

* Known coronary artery disease
* Renal Insufficiency(creatinine > 1.5 mg/dl)or renal failure requiring dialysis
* Pregnancy or unknown pregnancy status
* Clinical Instability as deemed by attending physician;including cardiogenic shock, sustained ventricular or atrial arrhythmia requiring intravenous medications, hypotension
* Patient's with known allergy to iodine or shellfish
* Inability to tolerate Beta Blockers
* Use of Viagra or Cialis in past 24 hours
* Body Mass (BMI)>38

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain over the age of 18 years old with symptoms of Coronary Artery Disease
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-03; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Raff, M.D., Study Director — Corewell Health East; James Goldstein, M.D., Study Chair — Corewell Health East; Michael Gallagher, M.D., Principal Investigator — Corewell Health East; Gilbert Raff, M.D., Principal Investigator — Corewell Health East